CLINICAL TRIAL: NCT01677065
Title: An Open-label, Single-dose, Randomized, Two-way Crossover Study to Estimate the Relative Bioavailability of a Controlled-release Formulation of Oxycodone (40 mg) With Sequestered Naltrexone Compared With Immediate-release Oxycodone Tablets (20 mg) in Healthy Volunteers
Brief Title: A Randomized, Two-way, Crossover Study to Estimate the Relative Bioavailability of a Controlled-release Formulation of Oxycodone (40 mg) With Sequestered Naltrexone Compared With Immediate-release Oxycodone Tablets (20 mg) in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B4531007; ALO-02 Bioavailability Study
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Bioavailability; Oxycodone; Healthy Volunteers
MeSH Terms: interventions — oxycodone naltrexone combination; Oxycodone

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment A: Controlled release oxycodone test formulation 40 mg
  Interventions: Drug: Oxycodone controlled-release test formulation
- Treatment B: Immediate release oxycodone reference drug 20 mg
  Interventions: Drug: Immediate-release reference drug

INTERVENTIONS:
Drug: Oxycodone controlled-release test formulation — single dose administration of test formulation under fasted conditions
  Other Names: ALO-02
  Groups: Treatment A
Drug: Immediate-release reference drug — single dose administration of reference drug under fasted conditions
  Other Names: Roxicodone
  Groups: Treatment B

SUMMARY:
To determine whether the bioavailability of the controlled-release test formulation is at least as high as that for the commercial reference drug.

DETAILED DESCRIPTION:
Serial sampling of venous blood

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers, greater than 50 kg, able and willing to sign informed consent

Exclusion Criteria:

* Evidence of significant illness, condition affecting drug absorption, history of sleep apnea, and allergy to opioid drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic endpoints - area under the concentration curve (AUC) | 0-48 hr

SECONDARY OUTCOMES:
Peak concentration (Cmax) and time to peak concentration (Tmax) | 0-48 hr

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4531007